CLINICAL TRIAL: NCT00373672
Title: Effect of Addition of Modafinil on the Tolerability and Efficacy for Cognition of Atypical Antipsychotic Drugs in Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Effects of Armodafinil on Cognition for Patients With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060567
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Armodafinil (Nuvigil) (Active Comparator): First group will be randomized to take Armodafinil (Nuvigil) 150 mg, along with their current anti psychotic medication and tested at baseline and week 6 for differences in memory, attention and problem-solving ability. Changes in weight during the six week study will also be tracked.
  Interventions: Drug: armodafinil (Nuvigil)
- Placebo (Placebo Comparator): Second group will be randomized to take placebo,identical in appearance to active comparator, along with their current anti psychotic medication and tested at baseline and week 6 for differences in memory, attention and problem-solving ability. Changes in weight during the six week study will also be tracked.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: armodafinil (Nuvigil) — armodafinil (Nuvigil)150 mg qd
  Arms: Armodafinil (Nuvigil)
Drug: placebo — identical in appearance to active comparator
  Arms: Placebo

SUMMARY:
This is a six week, double blind,placebo controlled study for patients with schizophrenia or schizoaffective disorder treated with an atypical antipsychotic for at least two months. Subjects will be randomized to take armodafinil (Nuvigil) or placebo along with their current antipsychotic and tested at baseline and week 6 for differences in memory, attention and problem-solving ability. Changes in weight during the six week study will also be tracked.

ELIGIBILITY:
Inclusion criteria

* Men and women age 18-65 years
* Patients with Diagnostic and Statistical Manual (DSM-IV) defined schizophrenia or schizoaffective disorder
* Treated with any atypical antipsychotic for at least 2 months
* Patients with documented weight gain > 7% with current antipsychotic medication
* Able to provide written consent

Exclusion criteria

* Women who are pregnant or nursing. Female participants must have a negative urine pregnancy test at screening.
* DSM-IV defined substance or alcohol dependence within the 2 months preceding the start of the trial
* Treatment with a monoamine oxidase inhibitor (e.g., tranylcypromine, phenelzine, isocarboxazid) within 2 weeks of starting the trial
* Patients considered at high risk for suicide or violence
* Patients with history of or symptoms on systems review consistent with clinically significant and currently relevant hematologic, renal, hepatic, gastrointestinal, endocrine, pulmonary, dermatologic, oncologic or neurologic (including seizures or epilepsy) disease
* Patients with a history of or symptoms on systems review consistent with significant cardiovascular disease, bypass surgery, or concurrent cardiovascular disease, including uncontrolled hypertension, hypotension, congestive heart failure, angina pectoris, or recent (within last 6 months) myocardial infarction
* Use of any investigational drug within 4 weeks before screening
* History of hypersensitivity or other intolerable adverse effects to modafinil
* Patients who experience severe sleep disturbances from modafinil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William V Bobo, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Bobo WV, Woodward ND, Sim MY, Jayathilake K, Meltzer HY. The effect of adjunctive armodafinil on cognitive performance and psychopathology in antipsychotic-treated patients with schizophrenia/schizoaffective disorder: a randomized, double-blind, placebo-controlled trial. Schizophr Res. 2011 Aug;130(1-3):106-13. doi: 10.1016/j.schres.2011.05.015. Epub 2011 Jun 8. PMID 21641776

RESULTS

PARTICIPANT FLOW:
Groups:
- ARM + APD: armodafinil (Nuvigil) 150 mg
  armodafinil (Nuvigil): armodafinil (Nuvigil)150 mg qd
- PLC + APD: identical in appearance to active comparator
  placebo: identical in appearance to active comparator
Period: Overall Study
Arm/Group | ARM + APD | PLC + APD
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM + APD | PLC + APD | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (14.6) | 38.8 (11.7) | 41.4 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 15 | 20 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Cognition Measured by AX-Continuous Performance Test (AX-CPT) D-prime Score
Description: For the AX-CPT, subjects are required to maintain an attentional set across a delay interval in order to overcome a prepotent response tendency (target responses are required when an X is presented but only in the context of a preceding A; non-target conditions are AY, BX and BY). The dependent measure was d-prime at the long delay (calculated as AX hits minus BX false alarms, which is particularly sensitive to context processing impairments in individuals with schizophrenia.
Time Frame: Baseline and week 6
Population: Treatment effects were analyzed using a repeated measures analysis of variance model with time (baseline, 6 weeks) as the within-subjects factor and treatment group (armodafinil, placebo) as the between-subjects factor.
Measure: Mean (Standard Error); unit: d prime score
Arm/Group | ARM + APD | PLC + APD
Number analyzed (Participants) | 29 | 29
d prime score
  Baseline | 2.7 (0.3) | 2.5 (0.3)
  6 weeks | 2.3 (0.4) | 3.2 (0.4)
Statistical Analysis 1: Comparison: ARM + APD vs PLC + APD; Treatment effects were analyzed using a repeated measures analysis of variance model with time (baseline, 6 weeks) as the within-subjects factor and treatment group (armodafinil, placebo) as the between-subjects factor; Test type: Superiority; p < 0.016, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | ARM + APD | PLC + APD
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 1/29 | 0/29
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM + APD (N=29) | PLC + APD (N=29)
worsening of psychiatric symptoms (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes